CLINICAL TRIAL: NCT01683864
Title: Randomized Controlled Trial to Prevent Peritoneal Seeding in Gastric Cancer
Acronym: HIPECStomach
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Recruitment problems
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-004405-25
Record Dates: First submitted 2012-09-06; First posted 2012-09-12 (Estimated); Results first posted 2018-01-30 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2016-10

CONDITIONS: Gastric Cancer; Peritoneal Carcinomatosis
MeSH Terms: conditions — Stomach Neoplasms; Peritoneal Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- positive cytology with HIPEC (Experimental): gastric cancer cytology positive with HIPEC Mytomycin and cisplatin intraoperative
  Interventions: Drug: positive cytology with HIPEC
- positive cytology without HIPEC (No Intervention): gastric cancer cytology positive without HIPEC
- negative cytology without HIPEC (No Intervention): gastric cancer with negative cytology

INTERVENTIONS:
Drug: positive cytology with HIPEC — HIPEC with mytomycin and cisplatin
  Other Names: mytomycin and cisplatin
  Arms: positive cytology with HIPEC

SUMMARY:
Randomized Controlled Trial to Prevent Peritoneal Seeding in Gastric Cancer

DETAILED DESCRIPTION:
The gastric carcinoma is one of the four most common tumors occurring worldwide. The advanced phase is characterized by metastasis and poses a very poor prognosis for survival. In 20%-30% of gastric carcinomas the tumor spreads into the abdominal cavity, which leads to metastases in the wall of the peritoneal cavity. This is known as peritoneal carcinomatosis and its five-year survival rate is less than 2%. Even after R0 resection of a localized gastric carcinoma the five-year survival rate is only 40%, not least of all because relapses in the form of peritoneal metastases are a common occurrence.

Patients with gastric carcinoma and not yet diagnosed with metastases, but who show free tumor cells in cytology in preoperative laparoscopy before neoadjuvant chemotherapy and gastrectomy, have an 80% risk of developing peritoneal carcinomatosis within one year, which stands in strong contrast to the 40% risk for patients with negative cytology.

In the study presented here (group A) therapeutic hyperthermic intraperitoneal chemoperfusion (HIPEC, in the literature also known as HIIC (heated intraoperative intraperitoneal chemotherapy) or IPHC (intraperitoneal chemohyperthermia)) with mitomycin c and cisplatin will be administered following gastrectomy in patients with a gastric carcinoma with free tumor cells in cytology diagnosed in the preoperative laparoscopy in comparison to (group B) solely gastrectomy in patients with a gastric carcinoma and also with free tumor cells diagnosed in cytology in the preoperative laparoscopy.

A randomization will be performed between group A and B. Patients with gastric carcinoma (TNM Stage ≥ T2<T4) without proven metastases (TNM stage M0), with and without involved regional lymph nodes (TNM stage +N/-N) and positive cytology in preoperative abdominal lavage will be included. Exclusion criteria are extended disease or inoperable tumor.

This study is already permitted by the local ethic commission and the German Federal Institute for Drugs and Medical Devices (BfArM) (EudraCT-Nr.: 2011-004405-25 / Study code: HIPEC_Stomach) and was initiated in August 2012.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven gastric adenocarcinoma: uT1,uT2, uT3, Nx, M0
2. No prior chemotherapy
3. Patients of full age, independent of gender ECOG ≤ 2
4. No dissemination of the tumor confirmed by CT of the lung and the abdomen.
5. Signed Consent form of the Patient agreeing to investigations
6. Leucocytes > 3.000/µl
7. Thrombocytes > 100.000/µl
8. Creatinine ≤ 1.5mg/dl and or Clearance > 60 ml/min
9. informed consent of the patient
10. normal ejection-fraction of the heart

Exclusion Criteria:

1. Dissemination of the tumor or non-resectable primary tumor
2. Malignant secondary disease < 5 years in the past (Exception: in-situ-carcinoma of the cervix and appropriately treated basal cell carcinoma of the skin)
3. Patient not of full age
4. Inflammatory chronic bowel disease
5. Inclusion of the patient in a different study
6. Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfred Königsrainer, MD, Principal Investigator — University Hospital Tuebingen
Locations (1):
- University of Tuebingen, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was early terminated due to recruitment problem. All active patient have study
Groups:
- Positive Cytology With HIPEC: gastric cancer cytology positive with HIPEC Mytomycin and cisplatin intraoperative positive cytology with HIPEC: HIPEC with mytomycin and cisplatin
Period: Overall Study
Arm/Group | Positive Cytology With HIPEC | Positive Cytology Without HIPEC | Negative Cytology Without HIPEC
Started | 0 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No study results because no patient has received study drug.
Groups:
- Positive Cytology no HIPEC: gastric cancer cytology positive without HIPEC
- Total: Total of all reporting groups
Arm/Group | Positive Cytology With HIPEC | Positive Cytology no HIPEC | Negative Cytology Without HIPEC | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0
Age, Categorical
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years |  |  |  | 0
  >=65 years |  |  |  | 0
Sex: Female, Male
  Female | 0 | 0 | 0 |

OUTCOME MEASURES:

1. Primary Outcome: Peritoneal Carcinosis Free Survival
Description: Three patients were enrolled in the study. No study results because no patient has received study drug.
Time Frame: 5 Years
Population: No study results because no patient has received study drug. Patient in the intervention group withdrawal of consent before intervention.
Groups:
- Positive Cytology With HIPEC: gastric Cancer cytology positive with HIPEC
- Positive Cytology Witout HIPEC: gastric cancer positive cytology without HIPC
- Negative Cytology Without HIPC: gastric cancer negative cytology without HIPC
Arm/Group | Positive Cytology With HIPEC | Positive Cytology Witout HIPEC | Negative Cytology Without HIPC
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Disease Free Survival
Description: No study results because no patient has received study drug.
Time Frame: 5 years
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Procedure Related Complication
Description: No study results because no patient has received study drug.
Time Frame: 60 days
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Kinetics of Mitomycin and Cisplatin
Time Frame: 24 hours after application
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- Positive Cytology With HIPEC: gastric cancer cytology positive with HIPEC Mytomycin and cisplatin intraoperative positive cytology with HIPEC: HIPEC with mytomycin and cisplatin Adverse Event : NA
- Positive Cytology no HIPEC: gastric cancer cytology positive without HIPEC Adverse Event : NA
- Negative Cytology Without HIPEC: gastric cancer with negative cytology Adverse Event : NA
Arm/Group | Positive Cytology With HIPEC | Positive Cytology no HIPEC | Negative Cytology Without HIPEC
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes